CLINICAL TRIAL: NCT01168570
Title: Progression of Renal Amyloidosis of FMF and Relation to Serum SAA Level
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba medical Center, Sheba Medical Center
Other Study IDs: SHEBA-10-7713-AL-CTIL
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Observational
Keywords: familial Mediterranean fever; amyloidosis AA; serum amyloid A; renal failure; nephrotic syndrome
MeSH Terms: conditions — Familial Mediterranean Fever; AA amyloidosis; Renal Insufficiency; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SAA monitored group: FMF-Amyloidosis patients receiving colchicine with a purpose to normalize SAA levels
- Historical control group: FMF-Amyloidosis patients receiving colchicine at a dose determined to stop FMF attacks. obtained from the Fibrillex study

SUMMARY:
Purpose of this study is to determine whether keeping SAA on normal or near normal level will delay progression of renal failure in patients with amyloidosis secondary to FMF.

DETAILED DESCRIPTION:
FMF is an inherited inflammatory disorder typically presented in most causes as recurrent episodes of fever and serositis. Phenotype II, another kind of this disorder, has atypical courses, when the inflammation proceeds without any clinical sign.

Each FMF attack is accompanied by sharp elevation of inflammatory markers in the serum, and serum amyloid A (SAA) one of them. The level of these inflammatory markers returns to normal with termination of the attack. The SAA is the main component of amyloids fibrils and constantly high level of SAA after the attack (as occurs in undiagnosed or undertreated disease) is the significant risk factor responsible for development of amyloidosis. On the other hand, in patients with phenotype II the amyloidosis occurs despite absolute absence of the attacks.

The kidney is one of the first organ suffers from amyloid deposits. The spectrum of kidney damage spread wildly from mild proteinuria to obvious nephrotic syndrome with disturbance in renal function and progression to end stage renal failure.

It is well known that deterioration of renal disease in AA amyloidosis links to level of SAA in serum. The permanently high SAA level is a major factor responsible to progression of renal disease. Occasionally, however, decline in the renal function occurred despite normal or near normal levels of SAA. Renal impairment in these cases may be explained by mechanisms existing in other kidney diseases when uncontrolled proteinuria aggravates renal dysfunction. The purpose of the study is to find whether a cohort of patients followed in our clinic and receiving colchicine for FMF- amyloidosis according to the SAA levels, monitored periodically, have better prognosis than an historical cohort receiving colchicine according to the attack status

ELIGIBILITY:
Inclusion Criteria:

* FMF patients with amyloidosis AA
* 18 year and older

Exclusion Criteria:

* patients with AA amyloidosis not related to FMF
* evidence of other primary renal disease or renovascular pathology
* evidence of renal disease secondary to any systemic illness
* presence of inflammatory, autoimmune conditions or chronic infection that could lead to high SAA level
* pregnancy
* inability to provide legal consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 FMF patients with AA amyloidosis demonstrated by positive biopsy of any target organs
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Avi Livneh, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Lachmann HJ, Goodman HJ, Gilbertson JA, Gallimore JR, Sabin CA, Gillmore JD, Hawkins PN. Natural history and outcome in systemic AA amyloidosis. N Engl J Med. 2007 Jun 7;356(23):2361-71. doi: 10.1056/NEJMoa070265. PMID 17554117
- [Background] Gillmore JD, Lovat LB, Persey MR, Pepys MB, Hawkins PN. Amyloid load and clinical outcome in AA amyloidosis in relation to circulating concentration of serum amyloid A protein. Lancet. 2001 Jul 7;358(9275):24-9. doi: 10.1016/S0140-6736(00)05252-1. PMID 11454373
- [Background] Yalcinkaya F, Cakar N, Acar B, Tutar E, Guriz H, Elhan AH, Ozturk S, Kansu A, Ince E, Atalay S, Girgin N, Dogru U, Aysev D, Ekim M. The value of the levels of acute phase reactants for the prediction of familial Mediterranean fever associated amyloidosis: a case control study. Rheumatol Int. 2007 Apr;27(6):517-22. doi: 10.1007/s00296-006-0265-6. Epub 2006 Nov 14. PMID 17103173